CLINICAL TRIAL: NCT03127995
Title: Multicenter Randomized Phase III Trial Comparing Hypofractionated Versus Standard Radiotherapy in Breast Cancer With an Indication for Regional Lymph Node Irradiation in Terms of Lymphedema Occurrence
Brief Title: Hypofractionated vs Standard Radiotherapy in Breast Cancer With an Indication for Regional Lymph Node Irradiation About Lymphedema Occurrence
Acronym: HYPOG-01
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: UNICANCER (Other)
Collaborators: National Cancer Institute, France (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: UC-0107/1604; 2016-A00702-49 (Other: Id-RCB)
Record Dates: First submitted 2016-12-15; First posted 2017-04-25 (Actual); Last update posted 2024-04-09 (Actual); Status verified 2024-04

CONDITIONS: Breast Cancer Female
Keywords: Breast Cancer pT1-3, pN0-N3, M0; Lymph Node Irradiation
MeSH Terms: interventions — Radiation Dose Hypofractionation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- HYPOFRACTIONATED (Experimental): 40 Gy / 15 fractions, 2.67 Gy per fraction, 5 fractions per week.
  If the patient is candidate for a boost it will be provided as follows:
  * sequential boost with 40 Gy to CTV breast in 15 fractions and 16 Gy to CTV boost in 8 fractions
  * or simultaneous integrated boost (SIB) with 42.3 Gy on CTV breast and 52.2 Gy on CTV boost in 18 fractions
  Interventions: Radiation: HYPOFRACTIONATED
- NORMOFRACTIONATED (Other): 50 Gy / 25 fractions, 2.0 Gy per fraction, 5 fractions per week.
  If the patient is candidate for a boost it will be provided as follows:
  * sequential boost with 50 Gy to CTV breast in 25 fractions and 16 Gy to CTV boost in 8 fractions
  * or simultaneous integrated boost (SIB) with 51.52 Gy on CTV breast and 63 Gy on CTV boost in 28 fractions
  Interventions: Radiation: NORMOFRACTIONATED

INTERVENTIONS:
Radiation: HYPOFRACTIONATED — 40 Gy/ 15 fractions / 3 weeks
  Other Names: Experimental Arm
  Arms: HYPOFRACTIONATED
Radiation: NORMOFRACTIONATED — 50 Gy/ 25 fractions / 5 weeks
  Other Names: Standard Arm
  Arms: NORMOFRACTIONATED

SUMMARY:
The standard treatment of localized breast cancers consists of surgical removal of the tumor at the breast or removal of the entire breast and lymph nodes (sentinel lymph node and / or axillary dissection) with or without chemotherapy followed by radiotherapy on the breast or thoracic wall and the lymph node areas from 5 to 6.5 weeks.

Shorter radiotherapy treatments over 3 weeks for breast cancer without lymph node involvement have been equally effective and have no more side effects in several clinical trials involving several thousand patients. This called hypofractionated radiotherapy has become a standard for breast cancers in the absence of lymph node involvement in postmenopausal women.

The objective of the HypoG01 trial is to evaluate hypofractionated radiotherapy in women who require radiotherapy in the breast or chest wall and lymph node areas by comparing standard over 5 to 6.5 weeks and hypofractionated irradiation over 3 weeks analyzing the possible side effects and in particular the risk of lymphedema (swelling of the arm on the side treated) and the effectiveness of these treatments

ELIGIBILITY:
Inclusion Criteria:

* Woman ≥ 18 years who had radical surgery for invasive breast cancer pT1-3, pN0-N3, M0 with either mastectomy or breast conservation. The patient can be included no matter the status of oestrogen receptor, progesterone receptor, malignancy grade, HER2 status.
* ECOG 0-2
* Axillary lymph node dissection of the axilla where the findings give indication for regional nodes radiotherapy to levels +/-I, +/- II, +/-III, +/-IV, +/-interpectoral nodes (Rötter) and +/-the IMN.
* Sentinel node biopsy documenting limited nodal disease without an indication for axillary lymph node dissection according to institutional, national or other trial guidelines are accepted.
* The patient may be a candidate for a boost to the tumour bed.
* Adjuvant systemic therapy with chemotherapy, endocrine therapy and anti-HER2 treatment is accepted.
* Neoadjuvant chemotherapy for downstaging according to institutional or national guidelines is accepted if there is not an indication for a boost in the area of regional nodes after surgery.
* Primary systemic therapy of an operable breast cancer is accepted.
* If the patient is not treated with chemotherapy, the patient must be randomized within 8 weeks from last surgery. If the patient has received adjuvant chemotherapy, the patient must be randomized within 4 weeks after the last series of adjuvant chemotherapy or within 42 days from last surgery in case of surgery after neoadjuvant or adjuvant chemotherapy.Breast implants are accepted.
* Connective tissue disease is allowed if the treating radiation oncologist finds radiotherapy indicated
* Postoperative infection and/or seroma giving indication for drainage during RT is accepted
* Women of childbearing potential must agree to use adequate contraception for the duration of study participation and up to 3 months following completion of therapy
* Signed informed consent
* Affiliated to the Social Security system

Exclusion Criteria:

* Previous breast cancer or DCIS of the breast.
* Bilateral breast cancer
* Patient with previous non-breast malignancy with the exception of cancer in complete remission for over 5 years and low risk of recurrence. Patients with the following diseases can be accepted despite less than 5 years disease free interval: carcinoma in situ of the cervix, melanoma in situ, basal cell carcinoma of the skin, squamous cell carcinoma of the skin
* The patient has an indication for boost to 1 or more regional nodes
* Previous radiotherapy to the chest region
* Patient enrolled in another therapeutic trial. Observational cohorts are accepted if the collection of data does not interfere with the current trial
* Pregnant or lactating
* Conditions indicating that the patient cannot go through the radiation therapy or follow up, or a condition where the treating radiation oncologist thinks the patient should not participate in the trial for example due to language problems.

Ages: 18 Years to 85 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1265 (Actual)
Dates: Start 2016-09; Primary Completion 2022-12-31 (Actual); Study Completion 2030-09 (Estimated)

PRIMARY OUTCOMES:
Arm Lymphedema | At 3 years
  Occurrence radiation-induced late morbidity measured as lymphedema of the arm on the treated side at 3 years after adjuvant radiotherapy as follows: At least≥ 10% increased arm circumference measured 15 cm proximal and/or 10 cm distal of the olecranon of the treated side relative to the baseline value, compared to the contralateral side circumference also relative to its baseline value.

SECONDARY OUTCOMES:
Functional Assessment | Before treatment, week 3 or week 7 of treatment according the treatment arm and boost realization, 6 months after the last fraction received, every year during 5 years, 10 years
  Flexion/abduction of the upper arm will be assessed.
Aesthetics Assessment-FIBROSIS | Before treatment, week 3 or week 7 of treatment according the treatment arm and boost realization, 6 months after the last fraction received, every year during 5 years, 10 years
  Fibrosis as tissue induration, telangiectasia, oedema of the breast/chest wall and dyspigmentation will be evaluated according the LENT-SOMA scoring scale.
Aesthetics Assessment-BIS SCORE | Before treatment, week 3 or week 7 of treatment according the treatment arm and boost realization, 6 months after the last fraction received, every year during 5 years, 10 years
  The patient evaluates satisfaction on The Body Image Score (BIS) where has been added an extra question regarding clothing habits and furthermore based on the study by Lyngholm et al also 2 more questions regarding the satisfaction with the appearance of the treated breast after breast conservation with and without comparison to the opposite breast as done in the DBCG HYPOII trial. In addition, it will ask if the patient treated with breast conservation has had lipo-feeling injection in the breast during follow up.
Aesthetics Assessment-Global Cosmestic | Before treatment, week 3 or week 7 of treatment according the treatment arm and boost realization, 6 months after the last fraction received, every year during 5 years, 10 years
  The global cosmetic result after breast conservation will be based on Harris´ 4-point scale modified by Rune Gärtner et al
CTCAE Toxicity Assessment | Before treatment, every week of treatment, week 3 or week 7 of treatment according the treatment arm and boost realization, 6 months after the last fraction received, every year during 5 years, 10 years
  Acute/ late toxicity will be assessed according to the flowchart and performed based on CTCAE V4
RTOG/EORTC Toxicity Assessment | Before treatment, every week of treatment, week 3 or week 7 of treatment according the treatment arm and boost realization, 6 months after the last fraction received, every year during 5 years, 10 years
  Acute/ late toxicity will be assessed according to the flowchart and performed based on Toxicity Criteria of RTOG/EORTC
Cancer Related events | 6 months after the last fraction received, every year during 5 years, 10 years
  Cancer related endpoints are secondary endpoints in this trial. It's a composite outcome taking into account all relapse events (locoregional, invasive disease, distant disease), breast-cancer specific survival, and causes of death as defined per DATECAN guidelines. All time to cancer related endpoints are defined as starting from the date of randomization until the event.
Cost-Utility | Week 3 or week 7 of treatment according the treatment arm and boost realization
  A cost-utility analysis comparing radiotherapy regimens will be performed based on QALYs
Quality of Life QLQ-C30 | Before treatment, week 3 or week 7 of treatment according the treatment arm and boost realization, 6 months after the last fraction received, every year during 5 years, 10 years
  Patients' quality of life will be assessed using self-administered questionnaire EORTC QLQ-C30
Quality of Life EORTC BR23 | Before treatment, week 3 or week 7 of treatment according the treatment arm and boost realization, 6 months after the last fraction received, every year during 5 years, 10 years
  Patients' quality of life will be assessed using self-administered questionnaire EORTC BR23
Quality of Life Euroqol EQ-5D5D | Before treatment, week 3 or week 7 of treatment according the treatment arm and boost realization, 6 months after the last fraction received, every year during 5 years, 10 years
  Patients' quality of life will be assessed using self-administered questionnaire Euroqol EQ-5D5D

CONTACTS AND LOCATIONS:
Overall Officials: Sofia RIVERA, M.D, Ph.D, Principal Investigator — Gustave Roussy, Cancer Campus, Grand Paris
Locations (28):
- France (28):
  - Clinique de l'Europe, Amiens
  - Institut de Cancerologie de L'Ouest-Paul Papin, Angers
  - Hôpital Jean Minjoz, Besançon
  - Institut Bergonie, Bordeaux
  - Centre Jean Perrin, Clermont-Ferrand
  - Hoptal Henri Mondor, Créteil
  - Centre Georges Francois Leclerc, Dijon
  - Centre Guillaume Le Conquerant, Le Havre
  - Centre de radiothérapie Hartmann, Levallois-Perret
  - Centre Galilée - Hôpital Privé La Louvière, Lille
  - Centre Oscar Lambret, Lille
  - Clinique Chenieux, Limoges
  - Hôpital du Scorff, Lorient
  - Centre Leon Berard, Lyon
  - Institut Paoli Calmettes, Marseille
  - ICM Val d'Aurelle, Montpellier
  - Institut de Cancerologie de Lorraine, Nancy
  - Centre Antoine Lacassagne, Nice
  - Hopital Saint-Louis, Paris
  - Institut Curie, Paris
  - Centre Eugene Marquis, Rennes
  - Centre Henri Becquerel, Rouen
  - Institut Curie- Rene Huguenin, Saint-Cloud
  - Institut de Cancerologie de L'Ouest-Rene Gauducheau, Saint-Herblain
  - Centre Paul Strauss, Strasbourg
  - Institut Claudius Regaud, Toulouse
  - CHU Bretonneau, Tours
  - Gustave Roussy, Villejuif

IPD SHARING:
Plan to Share IPD: Undecided